CLINICAL TRIAL: NCT02871830
Title: Effects of a Peer-led Walking In ScHools Intervention on Physical Activity Levels of Adolescent Girls: a School-based Cluster Randomised Controlled Trial
Brief Title: Effects of a Peer-led Walking In ScHools Intervention
Acronym: WISH project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REC/11/0236
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Physical Activity
Keywords: Physical activity; Walking; Intervention; Adolescent girls; Randomised trial
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention group (Experimental)
  Interventions: Behavioral: Physical Activity
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Physical Activity — 15 mins physical activity per day within the school setting.
  Arms: Physical activity intervention group

SUMMARY:
Children and young people are recommended to undertake at least 60 minutes of moderate to vigorous intensity physical activity each day. However recent findings have indicated that only 51% of children aged 7 years were meeting these guidelines. Previous research has also highlighted girls are significantly less active than. Furthermore, children living in Northern Ireland are least likely to meet the guidelines, with only 43.4% of children here reaching the recommended ≥ 60 minutes a day. The development of interventions which can successfully increase levels of physical activity in adolescent girls in Northern Ireland is of key importance. The aim of this intervention is to investigate whether or not girls (aged 11-13 years) can increase their daily levels of physical activity over a 12 week period by taking part in a school-based brisk walking intervention. The impact of participating in a school-based brisk walking intervention on a range of other outcome measures will also be investigated. A total sample of 200 adolescent females will be recruited onto the study, with recruitment of participants taking place at the school level. Following written consent from parents/guardians and assent from participants, participants will be randomised at the school level to either participate in the walking intervention or to act as controls. Objective physical activity will be assessed at 3 time points using an Actigraph accelerometer. At baseline, post-intervention (12 weeks) and follow up (4 months post-intervention) participants will also undergo measurements of height, weight, waist and hip circumference, bloody pressure, and cardiorespiratory fitness. Participants will also complete questionnaires assessing levels of physical activity and a number of psychosocial variables at each time point. Following completion of follow up measurements, a sub-sample of participants (n=45) will be invited to take part in focus groups to evaluate their experiences of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 11-13 years old
* Female
* Attend a school selected to take part in the study
* Healthy and free from any medical condition that limits their participation in a brisk walking intervention, for example, a musculoskeletal injury

Exclusion Criteria:

* Male pupils
* Those who are unable to walk or for whom walking is contraindicated will not be eligible for inclusion

Ages: 11 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Total daily physical activity | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Measured for 7 consecutive days using Actigraph accelerometer at each time-point

SECONDARY OUTCOMES:
Physical activity intensity | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Measured for 7 consecutive days using Actigraph accelerometer at each time-point
Self-reported physical activity | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Measured using Physical Activity Questionnaire for children
Weight | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
Blood pressure | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
Cardiorespiratory fitness | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Measured using the Queens College Step test
Self-efficacy for physical activity | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Psychosocial questionnaire - Children's physical activity self-efficacy scale
Self-efficacy for walking | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Psychosocial questionnaire - adapted walking self-efficacy scale
Social support for physical activity and walking | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Social support for physical activity and walking from male and female parents/guardians and friends scale
Attitude to exercise | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention
  Psychosocial questionnaire - perceived benefits and barriers to exercise scale
Waist hip ratio | Change between baseline and post-intervention (12 weeks) and 4-months post-intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlin A, Murphy MH, Nevill A, Gallagher AM. Effects of a peer-led Walking In ScHools intervention (the WISH study) on physical activity levels of adolescent girls: a cluster randomised pilot study. Trials. 2018 Jan 11;19(1):31. doi: 10.1186/s13063-017-2415-4. PMID 29325578